CLINICAL TRIAL: NCT06741748
Title: A Pragmatic, Multi-centre, Double-blinded, Two-arm Randomized Controlled Trial on a Direct Warming Frozen Embryo Transfer in Assisted Reproductive Technologies Treatment Outcome
Brief Title: Direct Warming Frozen Embryo Transfer Outcomes in Assisted Reproductive Technology
Acronym: DW-FET-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yiu Leung David Chan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.132-T
Record Dates: First submitted 2024-11-19; First posted 2024-12-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Frozen Embryo Transfer (FET); Assisted Reproductive Techniques; In Vitro Fertilization (IVF); Cryopreservation of Embryos; Pregnancy Outcome After in Vitro Fertilization (IVF)
Keywords: Direct Warming Method; Frozen Embryo Transfer; Assisted Reproductive Technologies; Cryopreservation; Cost-effectiveness in ART; Embryo Warming; In Vitro Fertilization

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model where participants are randomized into two groups: one group will receive the novel direct warming method, and the other group will undergo the conventional multi-step thawing method. Both groups will be followed to compare clinical outcomes such as pregnancy rates, live birth rates, and cost-effectiveness.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this trial, participants and outcomes assessors will be masked to ensure unbiased results. The embryologists performing the thawing procedures will not be masked, as they are directly involved in applying the assigned thawing method (either the direct warming method or the conventional multi-step method). Additionally, the research staff responsible for enrolling participants will also remain blinded to group assignments to maintain allocation concealment. However, participants who are determined not to be pregnant after embryo transfer may be informed of their group assignment at that time. However, if a pregnancy is confirmed, participants will not be informed of their group assignment until after delivery or in the event of pregnancy loss.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Warming method (Experimental): The blastocyst designated for thawing will be placed in a pre-warmed, direct warming medium for one minute. Afterward, the embryo is transferred into an embryo culture medium within a time-lapse system, where it remains until the patient is ready for the embryo transfer procedure. This direct warming method significantly reduces the total procedure time to approximately 3 minutes, making it about ten times faster than the conventional multi-step thawing method.
  Interventions: Other: Direct Warming Method
- Conventional multi-step thawing method (Placebo Comparator): In the conventional multi-step thawing method, vitrified blastocysts are sequentially thawed using a series of pre-warmed thawing, dilution, and washing solutions. The blastocyst is first placed in a thawing solution for 1-3 minutes, followed by immersion in a dilution solution for 4-6 minutes to reduce cryoprotectant concentration. Finally, the blastocyst is transferred to a washing solution for 5-10 minutes for rehydration. The entire process takes approximately 30 minutes, after which the embryo is placed into an embryo culture medium in a time-lapse system until it is ready for embryo transfer.
  Interventions: Other: Conventional Multi-step Thawing Method

INTERVENTIONS:
Other: Direct Warming Method — This intervention involves thawing vitrified blastocysts using a simplified, one-step direct warming method. The blastocyst is placed in a pre-warmed embryo culture medium for approximately one minute, then transferred directly into the embryo culture medium within a time-lapse system until ready for uterine transfer. The total thawing process takes approximately three minutes, reducing the duration and complexity of the procedure compared to conventional methods.
  Other Names: One-step thawing
  Arms: Direct Warming method
Other: Conventional Multi-step Thawing Method — This intervention involves thawing vitrified blastocysts using a standard, multi-step process. The procedure includes sequential exposure of the blastocyst to different thawing solutions containing varying concentrations of cryoprotectants, followed by its transfer into an embryo culture medium in a time-lapse system. The overall process takes approximately 10-30 minutes.
  Arms: Conventional multi-step thawing method

SUMMARY:
The goal of this clinical trial is to evaluate whether the direct warming method for frozen embryo transfers (FET) can improve live birth and pregnancy outcomes in women aged 18-45 undergoing IVF treatments. The main questions it aims to answer are:

* Does the direct warming method achieve a similar or higher clinical success rate for FET compared to the conventional multi-step method?
* Is the direct warming method more cost-effective than the conventional method?

Researchers will compare the direct warming method to the conventional multi-step method to see if the former leads to better pregnancy outcomes and reduced procedural time.

Participants will:

* Undergo either the one-step or conventional embryo thawing procedure.
* Complete standard clinical follow-ups for pregnancy, including ultrasound scans and pregnancy tests.

DETAILED DESCRIPTION:
This clinical trial explores a novel direct warming method for frozen embryo transfer (FET), aimed at improving both clinical and operational outcomes in assisted reproductive technologies (ART). The method was designed to simplify and accelerate the embryo thawing process, reducing the time needed for thawing while eliminating the use of cryoprotectants commonly required in conventional thawing methods. This innovation has the potential to offer a more efficient and cost-effective alternative to standard FET procedures.

The primary focus of this trial is to compare the clinical effectiveness of the direct warming method against the conventional multi-step thawing process. In particular, the study seeks to determine whether the new method yields comparable or superior outcomes in terms of clinical pregnancy rate (CPR), ongoing pregnancy rate (OPR), and live birth rate (LBR), while also assessing its overall cost-effectiveness.

Study Design and Technical Details

This study employs a randomized controlled design, with participants being allocated into either the intervention group (direct warming method) or the control group (conventional multi-step thawing). The direct warming method streamlines the thawing process to just 3 minutes, in contrast to the conventional method, which requires multiple stages and takes approximately 20 minutes. By using only an embryo culture medium without cryoprotectants, the direct warming method reduces both complexity and potential risks associated with handling and cryoprotectant toxicity.

Key Objectives

* Primary Objective: To evaluate the clinical efficacy of the direct warming method in achieving comparable or higher success rates for FET as compared to conventional multi-step thawing.
* Secondary Objective: To assess the cost-effectiveness of the direct warming method by comparing the consumable and time costs across different centers.

Expected Impact and Innovation

The direct warming method challenges the traditional multi-step thawing approach, offering a faster and simpler alternative without compromising clinical outcomes. By minimizing the need for cryoprotectants and reducing the complexity of the thawing process, the new method is expected to enhance the overall efficiency of FET procedures while maintaining or improving pregnancy success rates. Additionally, the cost and time savings associated with the direct warming method may make it a viable option for IVF clinics worldwide, driving standardization and consistency across clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Plan to undergo single embryo transfer (SET) during the FET cycle.
* Age between 18 and 45 years.
* Patients with at least one high-quality blastocyst available for transfer.
* Patients who have provided informed consent to participate in the study.

Exclusion Criteria:

* Patients with repeated implantation failure (RIF) or recurrent miscarriage (RM).
* Patients with known uterine anomalies or significant uterine pathology (e.g., fibroids, polyps).
* Patients who are unwilling or unable to provide informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 578 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 6-8 weeks post embryo transfer
  Number of participants with at least one intrauterine gestational sac observed on ultrasound at 6-8 weeks of gestation following embryo transfer.
Ongoing Pregnancy Rate (OPR) | 12 weeks post embryo transfer
  Number of participants with a viable intrauterine pregnancy observed on ultrasound at 12 weeks of gestation.
Live Birth Rate (LBR) | At delivery, approximately 9 months post embryo transfer
  Number of participants who deliver a live infant after 24 weeks of gestation.
Cost-Effectiveness | At the end of the study, approximately 4 years.
  A comparative analysis of the total costs, including costs of consumables (e.g., warming mediums, storage devices) and staff labor hours, associated with the direct warming method compared to the conventional multi-step thawing method. Costs will be measured in USD and analyzed at the end of the study period.

SECONDARY OUTCOMES:
Subgroup Analysis of Warming Medium | Throughout the study period, approximately 4 years.
  Analysis of the clinical differences between brands of warming mediums assessing their impact on embryo survival rate.
Subgroup Analysis of Storage Devices | Throughout the study period, approximately 4 years.
  Analysis of the clinical differences between brands of Storage Devices assessing their impact on embryo survival rate.

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (2):
  - The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong SAR
  - The CUHK Medical centre, Shatin,NT, Hong Kong SAR
- The Homerton Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD will not be shared due to concerns regarding participant confidentiality and privacy. Additionally, the informed consent process did not include provisions for the sharing of individual-level data with third parties. Furthermore, local regulatory restrictions limit the ability to distribute sensitive health data outside the study team.

REFERENCES:
- [Background] Canosa S, Parmegiani L, Charrier L, Gennarelli G, Garello C, Granella F, Evangelista F, Monelli G, Guidetti D, Revelli A, Filicori M, Bongioanni F. Are commercial warming kits interchangeable for vitrified human blastocysts? Further evidence for the adoption of a Universal Warming protocol. J Assist Reprod Genet. 2022 Jan;39(1):67-73. doi: 10.1007/s10815-021-02364-1. Epub 2021 Nov 30. PMID 34845576
- [Background] Wang SF, Seifer DB. Age-related increase in live-birth rates of first frozen thaw embryo versus first fresh transfer in initial assisted reproductive technology cycles without PGT. Reprod Biol Endocrinol. 2024 Apr 13;22(1):42. doi: 10.1186/s12958-024-01210-0. PMID 38615016
- [Background] Parmegiani L, Beilby KH, Arnone A, Bernardi S, Maccarini AM, Nardi E, Cognigni GE, Filicori M. Testing the efficacy and efficiency of a single "universal warming protocol" for vitrified human embryos: prospective randomized controlled trial and retrospective longitudinal cohort study. J Assist Reprod Genet. 2018 Oct;35(10):1887-1895. doi: 10.1007/s10815-018-1276-4. Epub 2018 Aug 3. PMID 30074129
- [Background] Schiewe MC, Anderson RE. Vitrification: the pioneering past to current trends and perspectives of cryopreserving human embryos, gametes and reproductive tissue. Journal of Biorepository Science for Applied Medicine. 2017;5:57-68.
- [Background] Jiang VS, Cherouveim P, Naert MN, Dimitriadis I, Souter I, Bormann CL. Live birth outcomes following single-step blastocyst warming technique - optimizing efficiency without impacting live birth rates. J Assist Reprod Genet. 2024 May;41(5):1193-1202. doi: 10.1007/s10815-024-03069-x. Epub 2024 Mar 13. PMID 38472563
- [Background] Liebermann J, Hrvojevic K, Hirshfeld-Cytron J, Brohammer R, Wagner Y, Susralski A, Jasulaitis S, Chan S, Takhsh E, Uhler M. Fast and furious: pregnancy outcome with one-step rehydration in the warming protocol for human blastocysts. Reprod Biomed Online. 2024 Apr;48(4):103731. doi: 10.1016/j.rbmo.2023.103731. Epub 2023 Nov 23. PMID 38359734
- [Background] Manns JN, Katz S, Whelan J, Patrick JL, Holt T, Merline AM, et al. VALIDATION OF A NEW, ULTRA-FAST BLASTOCYST WARMING TECHNIQUE REDUCES WARMING TIMES TO 1 MIN AND YIELDS SIMILAR SURVIVAL AND RE-EXPANSION COMPARED TO BLASTOCYSTS WARMED USING A STANDARD METHOD. Fertility and Sterility.
- [Background] Yan G, Yao Y, Yang W, Lu L, Wang L, Zhao D, Zhao S. An all-37 degrees C thawing method improves the clinical outcomes of vitrified frozen-thawed embryo transfer: a retrospective study using a case-control matching analysis. Arch Gynecol Obstet. 2023 Jun;307(6):1991-1999. doi: 10.1007/s00404-023-07029-1. Epub 2023 Apr 12. PMID 37041370
- [Background] Rienzi L, Gracia C, Maggiulli R, LaBarbera AR, Kaser DJ, Ubaldi FM, Vanderpoel S, Racowsky C. Oocyte, embryo and blastocyst cryopreservation in ART: systematic review and meta-analysis comparing slow-freezing versus vitrification to produce evidence for the development of global guidance. Hum Reprod Update. 2017 Mar 1;23(2):139-155. doi: 10.1093/humupd/dmw038. PMID 27827818
- [Background] Trounson A, Mohr L. Human pregnancy following cryopreservation, thawing and transfer of an eight-cell embryo. Nature. 1983 Oct 20-26;305(5936):707-9. doi: 10.1038/305707a0. PMID 6633637